CLINICAL TRIAL: NCT04007640
Title: Early Stages of Pancreatic Cancer Associated With Obesity and Metabolic Syndrome: Prevention and Screening Tools - Imaging of Fatty Pancreas in Humans: Correlation With Pathological Analysis
Brief Title: Early Screening of Pancreatic Lesions : Development of New Imaging Tools
Acronym: PAIR-PANCREAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other); Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A02712-53
Record Dates: First submitted 2019-04-16; First posted 2019-07-05 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Pancreatic Cancer
Keywords: Obesity; Diabetes; metabolic syndrome; Magnetic Resonance imaging,; Pancreatic Cancer; preneoplastic lesions; acino-ductal metaplasia,
MeSH Terms: conditions — Pancreatic Neoplasms; Obesity; Diabetes Mellitus; Metabolic Syndrome | interventions — Magnetic Resonance Spectroscopy; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Volunteer patient (Other): 1st stage: To adjust the transducer, test and validate pancreatic MRI sequences on volunteers without history of known pancreatic disorders. Adjustment of MRI parameters is needed to optimize data acquisition, especially in obese patients. Moreover, an external material (transducer) has to be applied on the abdomen. The right position has to be tested and specified before stages 2 and 3 of the study. We aim to include volunteers without history of known pancreatic disorders for the Stage 1, meaning volunteers without personal history or symptoms suggesting pancreatic disorders.
  Interventions: Radiation: MRI
- Obese volunteers with indication for hepatic MRI (Other): 2nd stage: To validate and assess pancreatic MRI sequences on obese volunteers with indication for hepatic MRI , in relation with acceptable resolution and field of view criteria applicable to the typical anteroposterior diameters found in obese persons. For Magnetic Resonance Elastography (MRE), the amplitude setting of the MRE transducer will be adapted to the size of obese patients, in addition to the aforementioned adjustments to spatial resolution and field of view sizes. The effect of frequency on MRE data quality will be investigated. The effects of respiratory motion will be investigated; indeed in obese patients respiration amplitude is typically low and this enables to acquire data in free breathing mode over long periods of time, which offers more possibilities (notably in terms of averaging, spatial resolution, mechanical wave sampling rate) than when constraining acquisition parameters with a maximum breath hold time of less than 20s.
  Interventions: Radiation: MRI with additional sequences
- Obese patient (Other): 3rd stage: To assess the relevance of MRI to diagnose specific pancreatic lesions in obese patients validated at the microscopic level. We will analyze MRI of obese patients and non-obese patients with a planned pancreatic surgery. It will be possible to compare imaging with histology performed on resected parenchyma
  Interventions: Procedure: Left pancreatectomy or pancreaticoduodenectomy; Radiation: MRI with additional sequences
- Non obese patients (Other): 3rd stage: To assess the relevance of MRI to diagnose specific pancreatic lesions in obese patients validated at the microscopic level. We will analyze MRI of obese patients and non-obese patients with a planned pancreatic surgery. It will be possible to compare imaging with histology performed on resected parenchyma
  Interventions: Procedure: Left pancreatectomy or pancreaticoduodenectomy; Radiation: MRI with additional sequences
- Overweight patients (Other): 3rd stage: To assess the relevance of MRI to diagnose specific pancreatic lesions in obese patients validated at the microscopic level. We will analyze MRI of obese patients and non-obese patients with a planned pancreatic surgery. It will be possible to compare imaging with histology performed on resected parenchyma
  Interventions: Procedure: Left pancreatectomy or pancreaticoduodenectomy; Radiation: MRI with additional sequences

INTERVENTIONS:
Radiation: MRI with additional sequences — MRI with 15 min additional sequences to validate and assess pancreatic MRI sequences
  Arms: Obese volunteers with indication for hepatic MRI
Radiation: MRI — MRI with 15 min additional sequences to validate and assess pancreatic MRI sequences
  Arms: Volunteer patient
Procedure: Left pancreatectomy or pancreaticoduodenectomy — Histological analysis :
  Arms: Non obese patients; Obese patient; Overweight patients
Radiation: MRI with additional sequences — MRI with 15 min additional sequences to assess the relevance of MRI to diagnose specific pancreatic lesions in obese patients
  Arms: Non obese patients; Obese patient; Overweight patients

SUMMARY:
Obesity, diabetes and metabolic syndrome (MS) have all been associated with increase of pancreatic cancer (PK) risk. The precise role of obesity and diabetes and the pathways involved in the early oncogenic phases of PK associated with MS are not well known. The investigators hypothesize that it is possible to decipher this specific "fat-fibrosis-neoplastic sequence", to develop new imaging tools adapted to follow its progression, to test the benefit of treatments to slow this sequence and prevent the development of PK in obese and diabetic patients.This project is in line with a prevention strategy, by planning to understand the physiopathological pathways involved in MS leading to PK, to develop tools useful to screen early precancerous lesions in order to diagnose and treat patients at high risk, before cancer involvement.

This clinical trial is part of the INCA PAIR PANCREAS project : Early stages of pancreatic cancer associated with obesity and metabolic syndrome:

prevention and screening tools - Imaging of fatty pancreas in humans: correlation with pathological analysis, which includes 3 main coordinated objectives an in vitro approach an in vivo approach and this study (clinical approach).

DETAILED DESCRIPTION:
Translational approach with direct application to humans, to test specific imaging MRI sequences in obese patients.

Obesity and metabolic syndrome are a well-known risk factor of pancreatic cancer. Obesity is associated with about 30% increased risk in all studies, but the proportion of obese people varies considerably from one country to another. Therefore, the proportion of cancer attributable to obesity could range from 3% to 16%. Numerous epidemiological studies confirmed that obesity is a risk factor of pancreatic cancer in obese men and women (BMI, kg/m2≥30.0), with a relative risk estimated to 1.76 (95% CI, 0.90-3.45) and 1.70 (95% CI, 1.09-2.64), respectively. As previously demonstrated by partners 9 and 10, obesity is associated with fat pancreatic infiltration and precancerous lesions, such as PanIN lesions in humans. Pancreatic lesions such as adipose infiltration, iron deposits, extent of fibrosis, acino-ductal metaplasia and Pan-IN are involved in pancreatic oncogenesis.

The goal of this study is to be able to diagnose early precancerous states in patients, such as acino-ductal metaplasia (and also PanIN lesions which are more frequently observed in humans,) inflammatory process (iron deposits, fibrosis lesions) and adipose involvement in the context of obesity and metabolic syndrome. Investigators hypothesis is that specific MR imaging sequences, adapted from previous studies in rodents, could be a relevant tool to diagnose early pancreatic lesions and follow their evolution in the context of obesity and metabolic syndrome.

To this aim, the investigators will conduct a study to assess the relevance of MR imaging sequences to diagnose specific pancreatic lesions in obese patients, validated at the microscopic level. The investigators will analyze MR imaging of obese patients (BMI>30)/non obese patients (BMI<25) with a planned pancreatic surgery. It will be possible to compare imaging with histology performed on resected parenchyma. The investigators propose a proof-of-concept study aiming at assessing the relevance of specific MR imaging to diagnose early pancreatic lesions in humans and in obese patients especially. MR imaging will be performed in both obese and non obese patients with a planned pancreatic surgery in hospital to resect a benign lesion (such as neuroendocrine tumour or IPMN...). MRI are performed in the normal course of care; their sequences will be adapted for this study. It will be possible to compare imaging with histology of the resected parenchyma.

ELIGIBILITY:
Inclusion Criteria:

* 1st stage : Volunteers without history of known pancreatic disorders

  - Adults
* 2nd stage : Obese Volunteers

  * Adults with planned hepatic MRI
  * Obese (BMI ≥30)
* 3rd stage : Patients

  * Adults (aged 18-65 years) with a planned pancreatic surgery for benign pancreatic lesions (IPMN, cystic lesions or neuroendocrine tumors)
  * Obese (BMI≥30), overweight (25≤BMI≤29.9) or non-obese patients (18.5<BMI<24.9)

Exclusion Criteria:

For volunteers without history of known pancreatic disorders (1st stage):

- Symptoms or past medical history suggesting pancreatic disorders

For all participants (1st, 2nd and 3rd stages) :

* Patients with contraindication to MRI (pacemaker, claustrophobia…)
* Inability to undergo MRI due to weight excess
* Pregnant or breastfeeding woman
* Absence of free and informed consent
* Non affiliation to a social security regime or CMU
* Subject deprived of freedom, subject under a legal protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2023-10-27 (Estimated); Study Completion 2023-10-27 (Estimated)

PRIMARY OUTCOMES:
Quantitative MRI parameters | Day 1
  Pancreatic fat content
Quantitative MRI parameters | Day 1
  Diffusion coefficients (10-4 mm2/s)
Quantitative MRI parameters | Day 1
  transverse magnetization relaxation rate
Quantitative MRI parameters | Day 1
  longitudinal relaxation rate
Quantitative MRI parameters | Day 1
  visco-elastic parameters by measure of tissue stiffness (kPa)
fibroinflammatory lesions at histology in obese patients | 2 months
  % surface of fibrosis
fibroinflammatory lesions at histology in obese patients | 2 months
  % surface of acinoductal metaplasia
fibroinflammatory lesions at histology in obese patients | 2 months
  number of acinoductal metaplasia lesions

SECONDARY OUTCOMES:
Histologic parameters | 2 months
  % surface of fat pancreatic infiltration
Histologic parameters | 2 months
  % surface of iron deposit
Histologic parameters | 2 months
  % surface of fibrosis
Histologic parameters | 2 months
  % surface of acinoductal metaplasia
Histologic parameters | 2 months y
  number of PanIN lesions
MRI parameters | Day 1
  pancreatic fat content
MRI parameters | Day 1
  Diffusion coefficients (10-4 mm2/s)
MRI parameters | Day 1I
  transverse magnetization relaxation rate
MRI parameters | Day 1
  longitudinal magnetization relaxation rate
MRI parameters | Day 1
  visco-elastic parameters by measure of tissue stiffness (kPa)
Biomarkers of pathways activation measured by immunohistochemistry on resected pancreatic parenchyma | 2 months
  % expression of molecules involved in TGFb and orexin signaling
Biomarkers of pathways activation measured by immunohistochemistry on resected pancreatic parenchyma | 2 months
  % expression of the markers in inflammatory cells (CD8, IL6, Caspase, HNF6)
Biomarkers of pathways activation measured by immunohistochemistry on resected pancreatic parenchyma | 2 months
  % surface of acinoductal metaplasia
Biomarkers of pathways activation measured by immunohistochemistry on resected pancreatic parenchyma | 2 months
  % of stained cells

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided